CLINICAL TRIAL: NCT02517710
Title: Single-blinded Prospective Trial Comparing Quantitive Blood Loss, Operative Time, and Post Operative Pain Using Stratafix Barbed Suture in Cesarian Section to the Use of Traditional Suture Material
Brief Title: Study to Compare Suture Material in Closure of Uterine Incision in Cesarian Section
Acronym: Stratafix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelical Community Hospital, Lewisburg, PA (Other)
Collaborators: Russell J.Stankiewicz, MD (Unknown); Ob/GYN Associates of Evangelical Hospital (Unknown); The Commonwealth Medical College (Unknown); Nickolas Serniak, BS, MS 4 (Unknown); Neil Cooper, MS, MS 4 (Unknown); Jennifer L. MacDonald, PA (Unknown)
Responsible Party: Principal Investigator, Russell J. Stankiewicz, MD, Assistant Clinical professor OB/GYN, Family Medicine, The Commonwealth Medical College, Evangelical Community Hospital, Lewisburg, PA
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ECH/TCMC101
Record Dates: First submitted 2014-10-09; First posted 2015-08-07 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Hysterotomy Closure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Group of patients receiving standard hysterotomy closure with synthetic braided suture
  Interventions: Procedure: Stratafix synthetic barbed suture
- Stratfix (Experimental): group of patients having the hysterotomy incision closed with barbed synthetic suture. Time to closure, blood loss, and postoperative pain
  Interventions: Procedure: Stratafix synthetic barbed suture

INTERVENTIONS:
Procedure: Stratafix synthetic barbed suture — hysterotomy closure in Cesarian section

SUMMARY:
Prospective single blinded trial comparing standard synthetic suture material to a synthetic barbed suture in closure of uterine incision, during Cesarean section procedures.

DETAILED DESCRIPTION:
Cesarean section is one of the most common medical procedures women of child bearing age undergo, in the United States and the world. This trial is designed to provide information and possible recommendation as to suture material used during closure of the uterus during that procedure. Our intent is to provide data relating to time of uterine closure, blood loss, and post operative pain. These conclusions may provide substantiated recommendations as to self locking and tying suture material in the performance of cesarean section as related to readily available synthetic suture material, which has the need for standard suture knot placement.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing age undergoing primary or repeat cesarean section using regional anesthesia.

Exclusion Criteria:

* General Anesthesia
* Non-consent to participation

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Blood loss in closure with barbed synthetic suture | 2 days
  monitoring of preoperative and postoperative hemoglobin and hematcrit

SECONDARY OUTCOMES:
Post operative pain after cesarean secton | 3 days
  using visual analog pain scale, compare standard closure to barbed suture closure pain

OTHER OUTCOMES:
time to close uterine hysterotomy incision comparing standard and barbed suture | total time comparision of closure rates over course of study period (2 years)
  comparing time to closure hysterotomy incision of standard suture verse barbed suture

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelical Community Hospital, Lewisburg, Pennsylvania, United States